CLINICAL TRIAL: NCT07404085
Title: Epigenetic Priming to Enhance Cognitive Training Gains and Neuroplasticity in Middle-age and Older Adults With Past Depression or Bipolar Disorder (EPIC)
Brief Title: Epigenetic Enhancement of Cognitive Training in Aging Mood Disorder Populations
Acronym: EPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Kamilla Woznica Miskowiak, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-25020884; P-2025-18923 (Other: [Registry ID: Danish Data Protection Agency])
Record Dates: First submitted 2025-12-11; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Disorder (BD); Depression - Major Depressive Disorder; Cognitive Impairment
Keywords: Cognition; Cognitive impairment; Mood disorders; Cognitive decline; Neuroplasticity
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction; Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1/4: VR high intensity + sodium butyrate (Experimental): VR high intensity: Virtual reality Based Cognitive Remediation Therapy (VR-CRT). The cognitive remediation programme has a duration of three weeks and involves weekly virtual reality-based cognitive training sessions with a therapist accompanied by additional between session homework assignments consisting of cognitively challenging daily life tasks.
  In this arm, VR high intensity (VR-CRT) is combined with daily intake of HDACi sodium butyrate.
  Interventions: Behavioral: Virtual Reality-based cognitive remediation therapy (VR-CRT); Dietary Supplement: HDACi butyrate
- Group 2/4: VR high intensity + placebo (Active Comparator): VR high intensity (VR-CRT): Same as above.
  In this arm, VR high intensity (VR-CRT) is combined with placebo.
  Interventions: Behavioral: Virtual Reality-based cognitive remediation therapy (VR-CRT); Dietary Supplement: Placebo
- Group 3/4: VR low intensity + sodium butyrate (Sham Comparator): VR low intensity: A virtual reality-based control treatment (VR-CT). This alternate treatment programme also has a duration of three weeks and involves one weekly 2-hour session with a therapist.
  In this arm, VR-based control treatment (VR-CT) is combined with daily intake of HDACi sodium butyrate.
  Interventions: Behavioral: Virtual Reality-based control treatment (VR-CT); Dietary Supplement: HDACi butyrate
- Group 4/4: VR low intensity + placebo (Sham Comparator): VR low intensity (VR-CT): Same as above.
  In this arm, VR-based control treatment (VR-CT) is combined with placebo.
  Interventions: Behavioral: Virtual Reality-based control treatment (VR-CT); Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Virtual Reality-based cognitive remediation therapy (VR-CRT) — VR-CRT on 360° Meta Quest 2-software in which participants train cognitive abilities guided by a therapist. The platform includes three immersive scenarios: (1) a kitchen scenario focusing on planning and cooking a meal, (2) a supermarket scenario focusing on grocery shopping and (3) a restaurant scenario focusing on remembering names and personal information. The virtual reality training is supported by a psychoeducation program that focuses on application of learned cognitive strategies in daily life.
  Arms: Group 1/4: VR high intensity + sodium butyrate; Group 2/4: VR high intensity + placebo
Behavioral: Virtual Reality-based control treatment (VR-CT) — VR-CT: The virtual reality control training involves completing different virtual reality games that are available through the Meta Quest games store. The chosen games involve no direct training of cognitive abilities such as planning skills og strategic learning, but merely involves simple reaction time and interaction with an entertaining environment that is meaningful to the participant and gives the impression of training cognitive skills.
  Arms: Group 3/4: VR low intensity + sodium butyrate; Group 4/4: VR low intensity + placebo
Dietary Supplement: HDACi butyrate — Daily intake of sodium butyrate.
  Arms: Group 1/4: VR high intensity + sodium butyrate; Group 3/4: VR low intensity + sodium butyrate
Dietary Supplement: Placebo — Daily intake of placebo.
  Arms: Group 2/4: VR high intensity + placebo; Group 4/4: VR low intensity + placebo

SUMMARY:
The aim of this clinical trial is to investigate the effects of a three-week virtual reality-based cognitive remediation training (VR-CRT) programme in combination with daily intake of a histone deacetylase inhibitor (HDACi) sodium butyrate on cognition in symptomatically stable patients with mood disorders (depression or bipolar disorder).

The investigators hypothesize that the VR-based cognitive remediation training (VR-CRT) combined with HDACi butyrate vs. a VR-based control treatment combined with placebo will improve global cognition (primary outcome measure) over three weeks.

Secondly, the investigators hypothesize that VR-CRT with placebo will improve cognition relative to the VR control treatment with placebo, although to a lesser extent than VR-CRT with HDACi butyrate.

Thirdly, the investigators hypothesize that the HDACi butyrate with VR control treatment will not produce cognitive improvements relative to placebo with VR control treatment.

Finally, the investigators hypothesize that the combined treatment (VR-CRT + HDACi butyrate) will enhance neuroplasticity (exploratory outcome) vs. VR control with placebo, as indicated by increase in hippocampal volume and/or memory-related activity shown with structural and functional MRI.

DETAILED DESCRIPTION:
The present study will include middle-age to older (40-75) outpatients with mood disorders (major depressive disorder or bipolar disorder) in full or partial remission (symptomatically stable) at the time of inclusion (≤ 14 on the Hamilton Depression Rating Scale - HDRS-17 or the Young Mania Rating Scale - YMRS). To accommodate an approximated drop-out rate of 15% from baseline to treatment completion (primary outcome assessment time point), the investigators will recruit up to 160 participants until full data sets are obtained for 120 participants (30 participants per arm).

Recruitment will be carried out through the outpatient Copenhagen Affective Disorder Clinic, other mental health centers in the Capital Region of Denmark, through consultant psychiatrists in the Capital Region and through advertisements on relevant websites.

After inclusion, baseline assessments are scheduled and completed over two days, one to five days apart. Participants are assessed with a VR-based virtual cognition test (CAVIR), and a comprehensive neuropsychological cognitive test battery. Participants also complete questionnaires concerning subjective cognitive complaints, quality of life, and personality traits. Psychosocial functioning is assessed using a clinician-rated interview and a performance-based assessment. Finally, sleep quantity and quality in the past 3 days is recorded. Within +/- 3 days an fMRI scan is carried out encompassing a spatial working memory N-back task, a word encoding paradigm in which participants encode and recall words of typical household items, an affective picture encoding test, in which participants denote the orientation (left/right) of emotionally valent pictures (incidental encoding), resting state, and a structural scan. After the scan, participants are asked to recall the emotional pictures encoded during the scan.

The virtual reality cognition test, neuropsychological assessments, questionnaires, clinical symptom ratings, assessment of psychosocial functioning and fMRI scan are repeated within 2 weeks of treatment completion (primary outcome assessment time). All assessments but fMRI are repeated again 1 month (4 weeks) after treatment completion.

Block randomization is carried out using the automated randomization module in the online Research Electronic Data Capture (REDcap) system based on an uploaded blocked randomization list stratified by age (< or ≥ 60 years) and diagnosis (major depressive disorder or bipolar disorder).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ICD-10 diagnosis of BD or recurrent UD in partial, or full remission (Hamilton Depression Rating Scale-17 items and Young Mania Rating Scale scores ≤14)
* Subjective cognitive complaints (self-reported: COBRA ≥12) or objectively-verified cognitive impairment (measured using Screening for Cognitive Impairment in Psychiatry SCIP: total score or at least two subscores ≥ 0.5 SD below expected norms)
* Fluency in Danish language

Exclusion Criteria:

* Diagnosis of schizophrenia
* Neurological disorders (including dementia)
* Dyslexia
* Severe Physical illness
* Kidney disease
* Cardiovascular disease
* Diabetes
* Alcohol or substance abuse
* Previous severe head trauma
* History of epilepsy
* Pregnancy or breastfeeding
* BMI >30
* Bodyweight < 45kg
* Daily use of benzodiazepines > 22.5 mg. oxazepam or > 7.5 mg. diazepam per day
* Serum lithium levels > 0.8 mmol/L
* Received electroconvulsive therapy < 2 months prior to participation
* Hypertension (>140 systolic or > 90 diastolic mm Hg)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive composite measure | Baseline, week 4 (treatment completion. Primary outcome assessment time point) and week 8 (follow-up)
  A global composite score based on the neuropsychological test across several cognitive domains: the Rey Auditory Verbal Learning Test (RAVLT)66 (verbal learning and memory), WAIS-III Letter-Number Sequencing 67 and Spatial Working Memory Test (CANTAB, SWM) (working memory), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)68 Coding (psychomotor speed), phonemic fluency and One Touch Stockings of Cambridge (CANTAB69, OTS) (executive function), RBANS Digit Span Test and Rapid Visual Information Processing (CANTAB69 , RVP), (attention) and Emotion Recognition Task (CANTAB69, emotional processing). No score range. higher scores mean a better outcome.

SECONDARY OUTCOMES:
Verbal memory composite | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  A composite score of RAVLT based on three subtests: total recall, immediate recall, and delayed recall (verbal learning and memory). No score range. higher scores mean a better outcome.
Cognition Assessment in Virtual Reality (CAVIR) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  The total score on our newly developed virtual reality-based daily-life real-world functioning test, Cognition Assessment in Virtual Reality (CAVIR). CAVIR includes 5 tests of verbal memory, executive functions, processing speed, working memory and attention, respectively. No score range. higher scores mean a better outcome.
Functional Assessment Short Test (FAST) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  A semi-structured interview assessing level of psychosocial functioning. Score range 0-72. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Rey Auditory Verbal Learning Test | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Neuropsychological test assessing verbal memory. Outcomes include total recall (score range 0-75), immediate recall (score range 0-15), and delayed recall (score range 0-15). Higher scores mean a better outcome.
Wechsler Adult Intelligence Scale (WAIS)-III Letter-Number Sequencing | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Neuropsychological test assessing working memory. Score range 0-21. Higher scores mean a better outcome.
Spatial Working Memory Test from Cambridge Cognition (CANTAB) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Computerized neuropsychological test assessing working memory. Outcomes include errors (score range 0-153, higher scores mean a worse outcome) and strategy (score range 3-26, higher scores mean a worse outcome).
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Neuropsychological test assessing psychomotor speed. Score range 0-89. Higher scores mean a better outcome.
Verbal fluency with letters "S" and "D" | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Neuropsychological test assessing executive functions. No score range. Higher scores mean a better outcome.
One Touch Stockings of Cambridge (OTS) from Cambridge Cognition (CANTAB) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Computerized neuropsychological test assessing executive functions. Outcomes include mean choices to correct (no score range, low scores mean a better outcome), problems solved on first choice (score range 1-15, higher scores mean a better outcome) and latency to correct (no score range, higher scores mean a worse outcome).
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Digit Span Test | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Neuropsychological test assessing attention. Score range 0-16. Higher scores mean a better outcome.
Rapid Visual Information Processing from Cambridge Cognition (CANTAB) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Computerized neuropsychological test assessing attention. Outcomes include signal detection (score range 0-1, higher scores mean a better outcome), probability of hit (score range 0-1, higher scores mean a better outcome), total false alarms (score range 0-546, higher scores mean a worse outcome), and latency to correct (score range 100-1900, higher scores mean a worse outcome).
Emotion Recognition Task | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Computerized neuropsychological test assessing emotion recognition. Outcomes include reaction time (no score range, higher scores mean a worse outcome) and hit rate (score range 0-1, higher scores mean a better outcome).
Cognitive Complaints in Bipolar Disorder Rating Scale (COBRA) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Questionnaire on subjective cognitive complaints. Score range 0-48. Higher scores means worse outcome
Cognitive Difficulties in Everyday Life (CODEL) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Questionnaire on subjective cognitive complaints. Score range 0-48. Higher scores means worse outcome
Hamilton Depression Rating Scale (HDRS-17) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Rating inventory assessing depressive symptoms. Score range 0-52. Higher scores mean a worse outcome.
Young Mania Rating Scale (YMRS) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Rating inventory assessing (hypo)manic symptoms. Score range 0-60. Higher scores mean a worse outcome.
Assessment of Quality of Life (AQoL-8D) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Questionnaire assessing quality of life. Score range 33-176. Higher scores mean a worse outcome.
World Health Organization Quality of Life (WHOQOL-BREF) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Questionnaire assessing quality of life. Score range 26-130. Higher scores mean a better outcome.
Work and Social Adjustment Scale (WSAS) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Questionnaire assessing occupational functioning. Score range 0-40. Higher scores mean a worse outcome.
Sheehan's Disability Scale (SDS) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Questionnaire assessing everyday functioning. Score range 0-30. Higher scores mean a worse outcome.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 4 (treatment completion) and week 8 (follow-up)
  Questionnaire assessing quality of sleep. Score range 0-21. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla Woznica Miskowiak, DMSc, DPhil, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital; Julian Macoveanu, PhD, Study Director — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Neurocognition and Emotion Across Disorders (NEAD Brain Centre, Copenhagen Affective Disorder Research Centre (CADIC), Psychiatric Centre Copenhagen, Frederiksberg Hospital, Frederiksberg, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No